CLINICAL TRIAL: NCT01698671
Title: InterGard Synergy Post-Marketing Surveillance Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCV00010173
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Aortic Aneurysm, Abdominal; Occlusive Disease of Artery of Lower Extremity
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- InterGard Synergy Vascular Graft (Other)
  Interventions: Device: InterGard Synergy Vascular Graft

INTERVENTIONS:
Device: InterGard Synergy Vascular Graft

SUMMARY:
The purpose of the study is to assess the performance and safety of the InterGard Synergy vascular graft.

DETAILED DESCRIPTION:
Study of the device in patients with aneurysmal and occlusive disease of the abdominal aorta and peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring an InterGard Synergy Vascular Graft

Exclusion Criteria:

* Patients with contra-indications per InterGard Synergy Vascular Graft
* Patients with current graft infection
* Patients with a known allergy to collagen, triclosan or silver acetate
* Patients who require urgent or emergent surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Graft Patency and Complications | 6 months
  * Patency will be assessed by color-coded duplex ultrasound up to 6 months post implantation.
  * Complications including the occurrence of graft infections will be assessed up to post implantation.

SECONDARY OUTCOMES:
Mortality rate | 6 months
  Mortality rate will be assessed up to 6 months post implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Max Zegelman, MD, Principal Investigator — Krankenhaus Nordwest
Locations (3):
- Study Centers, Graz, Vienna, Austria
- Germany (2):
  - Study Centers, Frankfurt, Karlsruhe
  - Study Centers, Heidelberg, Hamburg, Hanau